CLINICAL TRIAL: NCT01118832
Title: Using High Resolution Function Imaging To Detect Melanoma and Dysplastic Nevi
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Johns Hopkins University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0868; R01CA161265-02 (NIH); NA_00016040 (Other: JHM IRB)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Melanoma
Keywords: Thermography
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
A novel infrared imaging tool to aid in the clinical detection of atypical pigmented lesions and melanoma is developed. Goals include evaluation of the utility of high-resolution infrared scanning of cutaneous lesions in the diagnosis of pigmented lesions and the identification of high-risk lesions and melanomas.

DETAILED DESCRIPTION:
This study uses a specific skin protocol to cool the skin and then measures the cutaneous thermal recovery to uniquely identify lesions that may be cancerous. Using computer models, the thermal signature is used to determine the size and shape of the lesions in question. In particular, this study seeks to add quantification analysis of high resolution thermal images of melanoma lesions to provide accurate early diagnostic capability with specific detail regarding size, shape and depth of the lesions. This information will be compared to biopsy results and surgical resection results.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the high-risk pigmented lesion clinic, who posses a pigmented lesion with a clinical indication for biopsy

Exclusion Criteria:

* None

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The subject population will be identified in the Department of Dermatology Pigmented Lesion Clinic at the Johns Hopkins Hospital Outpatient Center. Recruited patients will only comprise those requesting a cutaneous pigmented lesion removed or patients that are examined and found to have a pigmented lesion that is suspicious for malignancy at the time of their visit, and thus recommended to have a skin biopsy for diagnosis following the standard of care
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2010-06-29 (Actual); Study Completion 2012-02-20 (Actual)

PRIMARY OUTCOMES:
Ability to Detect of the melanoma lesions | up to 2 years
  Using activated cooling methods we are measuring skin surface temperature recovery of specific lesions and comparing them to biopsy results of the lesions in question.

SECONDARY OUTCOMES:
Measurement of thermal signatures of benign cutaneous lesions | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cila Herman, Dr-Ing., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] C HERMAN, THREE-DIMENSIONAL THERMAL IMAGING FOR THE DETECTION OF SKIN LESIONS AND OTHER NATURAL AND ABNORMAL CONDITIONS - WO Patent WO/2012/009,359, 2012
- [Result] Herman C. Emerging technologies for the detection of melanoma: achieving better outcomes. Clin Cosmet Investig Dermatol. 2012;5:195-212. doi: 10.2147/CCID.S27902. Epub 2012 Nov 12. PMID 23204850
- See also: Video article describing the melanoma scanner — http://www.jove.com/video/2679/quantitative-visualization-detection-skin-cancer-using-dynamic
- See also: Review article discussing emerging technologies for the detection of melanoma — http://www.dovepress.com/emerging-technologies-for-the-detection-of-melanoma-achieving-better-o-peer-reviewed-article-CCID